CLINICAL TRIAL: NCT00861536
Title: An Open, Multicenter, Randomised, Parallel Group Pilot Study to Investigate Two Different Polyclonal Rabbit Immunoglobulin Preparations for Safety and Efficacy:A Comparison of ATG-Fresenius S to Thymoglobulin in Prophylaxis for Immunological High Risk Patients Following Renal Transplantation
Brief Title: Comparison of ATG to Thymoglobuline in Renal Transplantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 82/06
Record Dates: First submitted 2009-03-12; First posted 2009-03-13 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Transplantation, Kidney
Keywords: risk factors; immunology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ATG Fresenius (Experimental)
  Interventions: Drug: ATG Fresenius
- Thymoglobuline Genzyme (Active Comparator)
  Interventions: Drug: Thymoglobuline Genzyme

INTERVENTIONS:
Drug: ATG Fresenius — Day 0: 9 mg/kg bw bolus Days 1-4: 3 mg/kg bw/d
  Arms: ATG Fresenius
Drug: Thymoglobuline Genzyme — Day 0-3: 1.5 mg/kg bw/d
  Arms: Thymoglobuline Genzyme

SUMMARY:
An open, multicenter, randomised, parallel group pilot study to investigate two different polyclonal rabbit immunoglobulin preparations for safety and efficacy: A comparison of ATG-Fresenius S to Thymoglobulin in prophylaxis for immunological high risk patients following renal transplantation. This non-inferiority trial shall demonstrate that ATG-Fresenius S is as efficacious as Thymoglobulin but has a better tolerance and fewer side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Recipients, who are at least 18 years or older and have a high immunological risk defined by:

   The presence of at least one donor-specific antibody (class I and/or II) detected and specified by flow-technology (FlowPRA and single antigen beads), which are
   * For class I below the threshold of detection of a current CDC T-cell-/ and B-cell cross-match
   * For class II below the threshold of detection of a current CDC B-cell cross-match.
2. Patient receives a renal allograft only.
3. Female patients of child bearing age agree to maintain effective birth control practice during the study.
4. Patient has been fully informed and has given written or independent person witnessed oral informed consent.

Exclusion Criteria:

1. Patient is pregnant or breastfeeding.
2. Patient has a low immunological risk constellation, defined by receiving a kidney from a HLA-identical related living donor.
3. Patient and donor have a positive T-cell crossmatch.
4. Patient and donor are ABO incompatible.
5. Patient with combined transplantation.
6. Age of donor >75 years.
7. Cold ischemia time >40 hours.
8. Patient has leucopenia, defined as having at transplantation less than 3000/mm3 leukocytes.
9. Patient has thrombocytopenia, defined as having at transplantation less than 75000/mm3 thrombocytes.
10. Patient is allergic or intolerant to ATG-Fresenius S, Thymoglobulin, steroids, Tacrolimus or MMF.
11. EBV risk constellation (recipient EBV negative and donor EBV positive).
12. Patient or donor is known to be HIV positive.
13. Patient has a liver disease, defined as continuously having ASAT (SGOT) and/or ALAT (SGPT) levels greater than 3fold of the upper value of the normal range of the investigational site during the past 28 days.
14. Patient with malignancy or history of malignancy <2 years, except non metastatic basal or squamous cell carcinoma of the skin that has been treated successfully.
15. Patient has uncontrolled concomitant infections and/or severe diarrhea, vomiting, or active peptic ulcer.
16. Patient is unlikely to comply with the visits schedule in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Adverse events | Daily

SECONDARY OUTCOMES:
Rejection | Daily
Graft function | Daily
Patient survival | Daily
Graft survival | Daily

CONTACTS AND LOCATIONS:
Overall Officials: Juerg Steiger, MD,Prof, Principal Investigator — University Hospital Basel, Transplantation Immunology and Nephrology
Locations (1):
- University Hospital Basel, Transplantation Immunology and Nephrology, Basel, Switzerland